CLINICAL TRIAL: NCT05361044
Title: Metabolomics Based Prediction Model for Liver Graft Viability During Normothermic Regional Perfusion in Donation After Circulatory Death
Brief Title: Liver Graft Viability Assessment During Normothermic Regional Perfusion
Acronym: MAASTR3BOLOMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL21_1179
Record Dates: First submitted 2022-04-22; First posted 2022-05-04 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Liver Transplant Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donnor of liver grafts (Other): Blood samples And liver biopsy taken from the donnor
  Interventions: Biological: Blood samples Donnor

INTERVENTIONS:
Biological: Blood samples Donnor — Additional samples will be preleved in the Normothermic Regional Reperfusion at 30 min, and blood sample will be collected at the end of the Normothermic Regional Reperfusion (4 samples of 5ml).

SUMMARY:
With the increasing shortage of available donor organs, liver transplantation from donation after circulatory death (DCD) has been established in many countries to offer a therapeutic strategy for patients with end-stage liver disease beyond standard donation after brain death (DBD). In France, a controlled DCD (cDCD) program based on the use of normothermic regional perfusion (NRP) during organ procurement has been successfully implemented since 2015. This program has since shown excellent post-transplant outcomes with one-year patient and graft survival rates >90%. However, owing to very strict donor and graft selection criteria nearly one third of all potential liver grafts were not transplanted because of presumed poor quality. Furthermore, survival in cDCD liver transplantation which did not adhere to the current selection criteria was significantly lower (68% vs 94%) compared to the highly selected population. Thus, to further expand selection criteria and reduce discard rates without compromising outcomes, there is an urgent need for novel objective methods to assess graft quality prior to transplantation.

Graft quality assessment prior to transplantation has been a key challenge in liver transplantation for decades and still today the decision to accept or decline a graft before transplantation relies for the most part on ''gut feeling" of the procurement or transplant team. Currently, selection criteria for cDCD in France are based on donor data, liver biopsy results and hepatocyte injury markers AST and ALT. While donor data are only indirect indicators of graft quality, liver graft biopsy are highly pathologist dependant and do not provide a dynamic assessment. Hepatocyte injury markers during normothermic perfusion have been shown to only have limited value in predicting post-transplant graft function. In addition, several recent studies have suggested a superior predictive value of specific biomarkers in the liver through metabolomics. There is growing evidence that dynamic graft preservation such as NRP may even allow a direct analysis of key injury metabolites within solid organ grafts.

During cDCD procurement, liver grafts are exposed to donor warm ischemia which in combination with static cold storage causes ischemia-reperfusion injury (IRI) of the graft during implantation in the recipient. IRI is directly correlated to detrimental post-transplant complications such as primary non function and ischemic cholangiopathy or even recipient death.

Studies in animal models have revealed that mitochondria play a major role in IR injury and several mitochondrial signature metabolites for example succinate have been identified in various solid organ grafts such as livers, hearts and kidneys. Based on these results, our team and others have recently identified the release of a small auto fluorescent molecular compound of the mitochondrial respiratory chain, Flavin Mononucleotide (FMN), during the early phase of hepatic I/R injury. Furthermore, FMN has been shown to serve as a surrogate marker for impaired cellular energy production of the liver graft prior to transplantation and enable accurate prediction of post-transplant liver graft viability. Given the natural fluorescence of FMN, a real time quantification method has been established allowing to rapidly assess viability of human liver grafts during the procurement process. Of note, a team from the United Kingdom has validated this real-time FMN quantification during NRP of cDCD liver grafts. Interestingly, since mitochondrial injury is a universal signature of graft injury during the transplant process, FMN has the potential to serve as viability marker in other solid organs such as hearts, lungs and kidneys.

In addition, metabolomics approach allow the identification and quantification of many metabolites in a biological system through the use of high-throughput analytical technologies. It can give valuable information about what has, is and will occured in a specific tissu. In Liver transplantation, efforts have focused on studying early event of IR which are known to influence long term outcomes. It is however a complex pathway involving numerous metabolites. Metabolomic is therefore gaining interst in field of LT because it can enlight underlying metabolic process occurring during organ preservation and can lead the way toward a better evaluation of graft quality.

Thus, this study aims at developing a robust bio-clinical prediction model of liver graft viability during NRP using in depth metabolomics of perfusate and tissue in combination with available donor and graft characteristics

ELIGIBILITY:
Inclusion Criteria:

* All cDCD liver grafts allocated to one of the study centers undergoing NRP and where procurement of any abdominal organ is initiated
* Procurement performed by one of the four transplant teams
* non opposition by the donor or his family to organ donation
* non opposition by the recipient to participate in the study
* All Adult recipients on the waiting list for liver transplantation elligible for a liver procured after circulatory death according to the Agence de la Biomedecine.

  * Recipient, aged at least 18 years and less than 66 years,
  * Awaiting a first transplantation,
  * Recipients considered not too sick to cope with post-reperfusion syndrome not ventilated, no inotropic agents ...)
  * No major surgical history and no portal vein thrombosis; To minimize cold and recipient ischemic time (anastomotic time), patients where the recipient hepatectomy was predicted to be difficult were excluded
  * With a MELD score ≤ 25
  * Patient has been duly informed and has consented. Although the results of transplantations after DCD have very clearly improved over the years, clear information for the recipient and the provision of informed consent both remain essential. This means making clear to the patient the risk of primary nonfunction as well as of ischemic cholangiopathy and early arterial thrombosis.

Exclusion Criteria:

-- cDCD procurement where NRP fails or is not initiated due to technical reasons

- Graft reallocation after procurement to a transplant team not included in the study

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Composit endpoint: Number of major liver graft-related adverse events (LGRAE) containing - Graft dysfunction or primary non-function - Non-anastomotic biliary structure - Arterial complications | Unitl the end of study, an average of 3 years
Identification and Semi Quantification of FMN during normothermic regional perfusion | Unitl the end of study, an average of 3 years
  Metabolomic evaluation of the graft including various markers of interest (FMN, hypoxanthine, succinate, xanthine, NADH) measured by sepctroscopy and mass spectrometry (LC-MS), during CRN.
Identification and Semi Quantification of Hypoxanthine during normothermic regional perfusion | Unitl the end of study, an average of 3 years
  measured by spectroscopy and mass spectrometry (LC-MS), during CRN.
Identification and Semi Quantification of succinate during normothermic regional perfusion | Unitl the end of study, an average of 3 years
  measured by spectroscopy and mass spectrometry (LC-MS), during CRN.
Identification and Quantification of xanthine during normothermic regional perfusion | Unitl the end of study, an average of 3 years
  measured by spectroscopy and mass spectrometry (LC-MS), during CRN.
Identification and Semi Quantification of NADH during normothermic regional perfusionn | Unitl the end of study, an average of 3 years
  measured by spectroscopy and mass spectrometry (LC-MS), during CRN.
Sensitivity and Specificity analysis of the FMN regarding the composit endpoint of outcome 1 | Unitl the end of study, an average of 3 years
Sensitivity and Specificity analysis of the hypoxanthine regarding the composit endpoint of outcome 1 | Unitl the end of study, an average of 3 years
Sensitivity and Specificity analysis of the succinate regarding the composit endpoint of outcome 1 | Unitl the end of study, an average of 3 years
Sensitivity and Specificity analysis of the xanthine regarding the composit endpoint of outcome 1 | Unitl the end of study, an average of 3 years
Sensitivity and Specificity analysis of the NADH regarding the composit endpoint of outcome 1 | Unitl the end of study, an average of 3 years

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Department of HPB surgery and liver transplantation, Clichy
  - Department of general surgery and liver transplantation, Croix-Rousse University Hospital 103 Boulevard de la Croix Rousse, Lyon
  - Department of HPB surgery and liver transplantation, Paris
  - Department of HPB and Digestive Surgery, Rennes

IPD SHARING:
Plan to Share IPD: No